CLINICAL TRIAL: NCT06883565
Title: Tertiary Lymphoid Structures Related Genes Predicting Prognosis in Clear Cell Renal Cell Carcinoma: a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Ding-Wei Ye (Other)
Responsible Party: Sponsor-Investigator, Ding-Wei Ye, Study Director, Fudan University
Organization: Fudan University (Other)
Other Study IDs: 20250313-1
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Carcinoma (RCC)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High tertiary lymphoid structure related score petients
- Low tertiary lymphoid structure related score petients

SUMMARY:
The purpose of this research was to uncover the prognostic significance of tertiary lymphoid structures related genes from ccRCC patients with respect to clinical characteristics and outcomes. This offers a novel perspective on selecting populations for prostate cancer immunotherapy in future scenarios.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with renal cell carcinoma

Exclusion Criteria:

* incomplete medical records, inadequate follow-up information, and confirmed non-prostatic acinar adenocarcinoma

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The purpose of this research was to uncover the prognostic significance of tertiary lymphoid structures related genes from ccRCC patients with respect to clinical characteristics and outcomes. This offers a novel perspective on selecting populations for prostate cancer immunotherapy in future scenarios.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Correlation between the high or low score of TLS(tertiary lymphoid structure) related gene model and clinical features | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China